CLINICAL TRIAL: NCT06690736
Title: Chemokine Receptor 4 PET/CT Imaging of CXCR4-Related Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University (Other)
Collaborators: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Shaobo Yao, PhD, Prof., Tianjin Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TJMUGH-02
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: CXCR4-related Disease; Tumor; Positron Emission Tomography; Metastasis
Keywords: PET/CT; Chemokine receptor 4; Pentixafor; Pentixather
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CXCR4 PET/CT Imaging (Experimental): Intravenous injection of one dose of 2-5 mCi 68Ga/18F-Pentixafor/Pentixather. Tracer doses of radiotracers will be used to image lesions by PET/CT
  Interventions: Diagnostic Test: CXCR4 PET/CT Imaging

INTERVENTIONS:
Diagnostic Test: CXCR4 PET/CT Imaging — Each subject receive a single intravenous injection of 68Ga/18F-Pentixafor/Pentixather, and undergo PET/CT imaging within the specificed time.
  Other Names: 68/18F-Pentixafor; 68/18F-Pentixather

SUMMARY:
To evaluate the potential usefulness of 68Ga/18F-Pentixafor/Pentixather positron emission tomography/computed tomography (PET/CT) for the diagnosis of primary and metastatic lesions in various CXCR4-related disease patients.

DETAILED DESCRIPTION:
Subjects with various CXCR4-related disease patients underwent 68Ga/18F-Pentixafor/Pentixather PET/CT either for an initial assessment or for recurrence detection. Lesions uptake was quantified by the maximum standard uptake value (SUVmax). The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and accuracy of 68Ga/18F-Pentixafor/Pentixather PET/CT were calculated.

ELIGIBILITY:
Inclusion Criteria:

* suspected or confirmed untreated Lymphoproliferative and other CXCR4-related diseases patients
* 18F-FDG PET/CT within two weeks
* signed written consent.

Exclusion Criteria:

* pregnancy
* breastfeeding
* known allergy against Pentixafor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value (SUV) | 30 days
  Standardized uptake value (SUV) of FAPI for each target lesion of subject or suspected primary tumor or/and metastasis.

SECONDARY OUTCOMES:
Diagnostic efficacy | 30 days
  The sensitivity, specificity and accuracy of FAPI PET/CT were calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No